CLINICAL TRIAL: NCT06190080
Title: Outcomes of Children With Eosinophilic Esophagitis: a Prospective Monocentric Observational Study
Brief Title: Outcome of Children With Eosinophilic Esophagitis
Acronym: Obs-OE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-HPNCL-05
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Esophagitis, Eosinophilic
Keywords: children; eosinophilic esophagitis; life quality
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management of eosinophilic esophagitis (Other): Follow-up visits are always organized in the same way. A consultation with a gastropediatrician will take place, with assessment of symptoms (PEESS score) and quality of life (PedsQL module for eosinophilic esophagitis and PedsQL 4.0 Generic Core Scales). Then, if treatment needs to be introduced or changed, a digestive endoscopy with biopsies will be carried out at 3 months to determine whether the patient is in remission or not. Depending on the results, the patient may be advised to adapt or maintain the current treatment.
  Interventions: Other: Digestive endoscopy

INTERVENTIONS:
Other: Digestive endoscopy — Digestive endoscopies are performed in the operative room under general anaesthetic 3 months after the introduction or change of treatment. Biopsies of the upper, middle and lower thirds of the esophagus will be taken and analyzed for pathology.

SUMMARY:
The investigator would like to create a prospective cohort of patients in order to describe eosinophilic esophagitis with the specificities corresponding to our geographical territory, and to study their evolution at 3 months, 6 months, 12 months, 18 months and 24 months.

This study would also enable us to investigate the quality of life of these chronically ill patients

DETAILED DESCRIPTION:
The investigator would like to create a prospective cohort of 16 patients included over 2 years in order to determine the rate of complete remission (clinical, endoscopic and histological) at 3 months, 6 months, 12 months, 18 months and 24 months of treatment initiation. It is also planned to describe this cohort of pediatric EO patients at inclusion and throughout follow-up, and to study their quality of life.

Follow-up visits is organized every 3 months with a gastropediatrician, who assesses the patient's symptoms (PEESS score) and quality of life (PedsQL eosinophilic esophagitis module and PedsQL 4.0 Generic Core Scales).

If treatment needs to be introduced or changed, a digestive endoscopy with biopsies will be carried out at 3 months to determine whether the patient is in remission or not.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OE according to the diagnostic criteria of the PNDS published in July 2022
* Due to start treatment.
* informed consent from one of the 2 parents or the representative of parental authority.
* Membership of a social security scheme.

Exclusion Criteria:

-

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of complete remission | at 3 months, 6 months, 12 months, 18 months and 24 months from treatment initiation.
  Complete remission will be defined according to the following criteria:
  1. Abolition of clinical symptoms as assessed by the Pediatric Eosinophilic Esophagitis Symptom Score
  2. Endoscopic score: EoE Endoscopic Reference Score (EREFS) ≤ 2 in the lower, middle and upper thirds of the esophagus.
  3. Eosinophilic infiltrate < 5/HPF in standard HES (Haemato-Eosin-Safran) stain on biopsies from lower, middle and upper thirds of esophagus
  4. No therapeutic change at follow-up visit to assess remission

SECONDARY OUTCOMES:
Description at inclusion of a cohort of pediatric patients with OE | throught a 24 months follow-up
  The description of the population will be carried out at baseline and during a 24 months follow-up at each consultation (M3, M6, M12, M18 and M24) by the patient's referring physician, listing :
  * demographic (age, gender, lifestyle) and medical (history, allergies, etc.) data at baseline only
  * Clinical data (types of symptoms, possible complications, etc.)
  * Paraclinical data (endoscopic and anapathic scores at diagnosis)
evolution of quality of life | at diagnosis, 3 months, 6 months, 12 months, 18 months and 24 months of treatment
  Quality of life will be measured using the Pediatric Quality of Life Questionnaire (PedsQL Eosinophilic Esophagitis part ) currently being validated in French by our team.
  The PedsQL eosinophilic eosophagitis module is divided into several forms, each corresponding to different age groups with questions adapted according to age. (2-4 years, 5-7 years, 8-12 years and 13-18 years). This questionnaire is intended for children and their parents.
  The total score is the sum of the 35 items for 8-17 year olds, 22 for 2-4 year olds, 27 for 5-7 year olds. The maximum score is 175 for 8-17 year olds, 110 for 2-4 year olds, 135 for 5-7 year olds. The higher the score, the greater the impact of eosinophilic esophagitis on the patient's life.
  Nevertheless, we will also use a more general quality-of-life questionnaire, the PedsQL 4.0 Generic Core Scales in its French version.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux pédiatriques de Nice CHU Lenval, Nice, France